CLINICAL TRIAL: NCT05440591
Title: Effects of Dapagliflozin and Metformin on Vascular Function in Newly-Diagnosed Treatment-Naive Type 2 Diabetes- A Randomised Controlled Trial (DMVascular Study)
Brief Title: Effects of Dapagliflozin and Metformin on Vascular Function in Newly-Diagnosed Treatment-Naive Type 2 Diabetes
Acronym: DMVascular
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tan Tock Seng Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DMV001
Record Dates: First submitted 2022-06-27; First posted 2022-07-01 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — dapagliflozin; Metformin; Tablets

STUDY DESIGN:
Intervention Model Description: Open Label Parallel Randomised Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Metformin (Active Comparator): Metformin XR 500 mg tablets - up-to twice daily orally.
  Interventions: Drug: MetFORMIN 500 Mg Oral Tablet
- Dapagliflozin (Experimental): Dapagliflozin 10 mg tablets - once daily
  Interventions: Drug: Dapagliflozin
- MetforminXR 500/Dapagliflozin 5mg (Experimental): MetforminXR 500/Dapagliflozin 5mg , tablets- once daily
  Interventions: Drug: Dapagliflozin / metFORMIN Pill

INTERVENTIONS:
Drug: Dapagliflozin — Dapagliflozin 10mg tablets
  Arms: Dapagliflozin
Drug: MetFORMIN 500 Mg Oral Tablet — Metformin 500 mg tablets twice daily
  Arms: Metformin
Drug: Dapagliflozin / metFORMIN Pill — Combination pill
  Arms: MetforminXR 500/Dapagliflozin 5mg

SUMMARY:
Trial Design: This is a 12 week randomised controlled open label trial comparing the impact of Dapagliflozin, Metformin and combination therapy on vascular function in newly diagnosed T2DM patients.

DETAILED DESCRIPTION:
Trial Design: This is a 12 week randomised controlled open label trial comparing the impact of Dapagliflozin, Metformin and combination therapy on vascular function in newly diagnosed T2DM patients.

Trial Participants: Approximately 150 newly diagnosed T2DM patients with randomization 1:1:1 to Metformin XR 500mg twice daily, Dapagliflozin 10 mg daily or Metformin XR 500/Dapagliflozin 5 mg daily

Primary Aim : To evaluate the influence of intervention on vascular function.

Secondary Aims:

1. To evaluate the influence on other parameters of vascular function and beds.
2. To evaluate the haemodynamics involving blood pressure regulation.
3. To evaluate the effects of SGLT2i versus Metformin on endothelial interactions (vascular permeability) and leukocyte-endothelial interactions (leukocyte rolling, adherence), endothelial regenerative capacity and other endothelial related pathways.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to give informed consent
2. Age 30-65 years
3. Newly diagnosed (within the past 1 - 2 years) to have T2DM and not started on diabetes medications, HbA1c 6.4% to 10% (both inclusive) and/or OGTT 0 min glucose ≥7.0mmol/L and/or 120 min glucose ≥11.8mmol/L OR Recently diagnosed to have T2DM and treated with Metformin for not more than 5 years, HbA1c ≤ 8%
4. No recent change in medications or new medications
5. eGFR>60mL/min/1.73m2
6. Patient is otherwise well with no acute systemic illness in the last 2 weeks.
7. Female participants of child bearing potential and male participants whose partner is of child bearing potential must be willing to ensure that they or their partner use effective contraception during the trial

Exclusion Criteria:

1. History of ketoacidosis or any other conditions causing acidosis e.g. Alcohol dependence
2. Has a history of urinary tract infections or is at risk for urinary tract infections (e.g prostatomegaly, vesicoureteric reflux, kidney stones)
3. Patients on corticosteroids or immunosuppressive agents
4. Patients known to have HIV infection and/or on anti-retroviral agents
5. Patients with typical clinical features suggestive of T1DM (young onset with no family history of diabetes or first presentation as DKA were excluded). The endocrinologist (PI or co-I) will look at the patient profile to confirm diagnosis of T2DM.
6. Has severe liver dysfunction
7. Considered inappropriate by investigators due to any other reason.
8. Female participant who is pregnant, lactating or planning pregnancy during the course of the trial.
9. Significant renal impairment.
10. Scheduled elective surgery or other procedures requiring general anaesthesia during the trial.
11. Participants who have participated in another research trial involving an investigational product in the past 12 weeks.
12. Participants who have a history of Peripheral Arterial Disease or peripheral vascular disease or complains of lower limb claudication pain.

    -

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2023-05-10 (Estimated); Study Completion 2023-05-10 (Estimated)

PRIMARY OUTCOMES:
Endothelial Function measured as reactive hyperaemia index (RHI-EndoPAT) | 3 months after initiation
Carotid Femoral Pulse Wave Velocity | 3 months after initiation
  Sphygmocor determined cf-PWV

SECONDARY OUTCOMES:
Augmentation index | 3 months after initiation
  Augmentation index-sphygmocor derived and RHI-endoPAT derived
Central pulse pressure | 3 months after initiation
  CPP-Sphygmocor derived
Advanced glycation end products | 3 months after initiation
  AGE reader measurements

CONTACTS AND LOCATIONS:
Overall Officials: Rinkoo Dalan, Principal Investigator — Tan Tock Seng Hospital
Locations (1):
- Tan Tock Seng Hospital, Singapore, Singapore